CLINICAL TRIAL: NCT01745016
Title: The Effect of 28 Days of Beta-alanine Supplementation on the Physical Working Capacity at Heart Rate Threshold (PWCHRT)
Brief Title: Effect of Beta-Alanine on Heart Rate Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Abbie Smith-Ryan, PhD, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: 12-1787
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Exercise; Fatigue
Keywords: dietary supplement; carnosine
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo
- Beta-Alanine (Experimental): beta-alanine
  Interventions: Dietary Supplement: Beta-alanine

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Beta-alanine
  Arms: Beta-Alanine

SUMMARY:
Beta-alanine, as a method to increase muscle carnosine, has been shown to enhance muscle buffering capacity and delay fatigue. Various fatigue tests have been utilized to examine the effectiveness of beta-alanine supplementation. The physical working capacity test has been used to show significant increases in physical working capacities following supplementation. The physical working capacity tests were originally developed by Moritani et al. 1981 and Devries et al. 1982 to measure the point of onset of muscular fatigue. It is hypothesized that beta-alanine will increase physical working capacity at heart rate threshold, thereby signifying a delay in fatigue.

DETAILED DESCRIPTION:
An equal number of men and women will be recruited [Men, n=20 (10 placebo [PL]; 10 beta-alanine (Active)]; [Women,n=20 (10 PL; 10 Active)]. Men and women will be randomly assigned to respective groups to allow for equal numbers in supplement and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35 years old
* Be recreationally active (defined as accumulating 1-5 hours of moderate intensity

Exclusion Criteria

* Any health risks or indicators that would prevent them from participating in physical activity, as determined by a health history questionnaire
* Must not have taken performance enhancing supplements containing beta-alanine or creatine during the last 3 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Physical working capacity at heart rate threshold | 0 to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Exercise and Sport Science, Chapel Hill, North Carolina, United States